CLINICAL TRIAL: NCT00851916
Title: VIRTUAL HDR CYBERKNIFE RADIOSURGERY FOR LOCALLY RECURRENT PROSTATIC CARCINOMA: A PHASE II STUDY
Brief Title: CyberKnife Radiosurgery for Locally Recurrent Prostate CA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CyberKnife Centers of San Diego (Other)
Responsible Party: Principal Investigator, Carlyn Tripp, Donald Fuller, M.D., CyberKnife Centers of San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CK Recurrent Prostate SD
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CyberKnife Radiosurgery (Other): Single arm study using CyberKnife radiosurgery to treat recurrent prostate cancer patients that have already received external beam radiotherapy.
  Interventions: Radiation: CyberKnife Radiosurgery

INTERVENTIONS:
Radiation: CyberKnife Radiosurgery — CyberKnife Radiosurgery

SUMMARY:
The purpose of this study is to scientifically evaluate the effects (good and bad) of a new type of radiation treatment in patients with locally recurrent prostate cancer after prior radiotherapy. The treatment is known as prostate radiosurgery, and is distinguished from traditional radiotherapy by the application of smaller, more precisely controlled margins around the area targeted for full dose radiation, and far fewer treatments, using a much larger dose per treatment.

This research is being done to see what advantages, if any, prostate radiosurgery may have over other salvage treatment methods, including brachytherapy, cryosurgery, high intensity focused ultrasound (HIFU), hormonal therapy and radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent adenocarcinoma of the prostate, clinical stage T1 - T3 (AJCC 6th Edition, see Appendix II), NX/N0, M0, following prior prostate radiotherapy.
* Karnofsky performance status >80.
* Greater than 5 year life expectancy
* Greater than 2 years since the original course of radiotherapy.
* Absence of distant metastases by radiologic or pathologic assessment.
* Absence of lymph node involvement by radiologic or pathologic assessment.
* Patients must sign a study-specific informed consent form prior to study entry.

Exclusion Criteria:

* Stage T4 disease (AJCC 6th Edition, see Appendix II).
* Less than 2 years since the original course of radiotherapy.
* Lymph node involvement (N1).
* Evidence of distant metastases (M1).
* Radical surgery for carcinoma of the prostate
* Previous or concurrent cancers other than basal, in situ, or squamous cell skin cancers unless disease-free for ≥ 5 years.
* Major medical or psychiatric illness, which in the investigator's opinion, would prevent completion of treatment and would interfere with follow-up.
* History of inflammatory bowel disease
* Late GI or GU Morbidity > Grade 1 from the prior course of radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-02; Primary Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Establish pattern of PSA decline | Post CyberKnife Radiosurgery - 5 year f/up

SECONDARY OUTCOMES:
Quality of Life realitive to other commonly used radiation treatment methods for recurrent prostate cancer | Post CyberKnife Radiosurgery/5 yr. f/up

CONTACTS AND LOCATIONS:
Overall Officials: Donald B Fuller, M.D., Principal Investigator — CyberKnife Centers of San Diego
Locations (1):
- CybeKnife Centers of San Diego, San Diego, California, United States